CLINICAL TRIAL: NCT05478460
Title: Acute and Chronic Pain After Video-assisted Thoracoscopic Surgery for Lung Cancer in Patients With Preoperative CT-guided Hookwire Localization
Brief Title: Acute and Chronic Pain After Video-assisted Thoracoscopic Surgery for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, chairman of Department of Anesthesiology, Fudan University
Other Study IDs: pain assessment after VATS
Record Dates: First submitted 2022-05-30; First posted 2022-07-28 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Video-assisted Thoracoscopic Surgery; hookwire location
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Before operation,patients were performed CT -guided hook wire localization(20G×120mm, PAJUNK medizintechnologie, Geisingen in Germany). patients were placed on a CT table in a suitable position(supine, prone, lateral) to obtain the shortest needle insertion route for their initial CT scan. Local anesthesia of the skin and planned puncture tract was performed using 10ml Lidocaine 1%. Next, the needle was inserted into or near the pulmonary nodule.
  Interventions: Other: Hookwire localization
- Group B: without hookwire localization

INTERVENTIONS:
Other: Hookwire localization — Patients were performed CT -guided hook wire localization(20G×120mm, PAJUNK medizintechnologie, Geisingen in Germany). patients were placed on a CT table in a suitable position(supine, prone, lateral) to obtain the shortest needle insertion route for their initial CT scan. Local anesthesia of the skin and planned puncture tract was performed using 10ml Lidocaine 1%. Next, the needle was inserted into or near the pulmonary nodule.
  Groups: Group A

SUMMARY:
The aim of this study is to evaluate whether preoperative CT- guided hookwire localization would influence the incidence and intensity of acute and chronic pain after VATS.

DETAILED DESCRIPTION:
Postoperative pain after thoracic surgery has gained recognition as a adverse outcome and head-scratching problem. The incidence of choric postoperative pain (CPSP) in thoracic surgery has been reported to be 20%-80%. However, there has been not an standard treatment for CPSP. Many study has showed the risk factors of CPSP in thoracic surgery, such as VATS type, operation time, duration of drainage, preoperative pain, repeat surgery, gender, postoperative chemotherapy or radiation therapy , etc. It is important that moderate-to-severe acute postoperative pain will be transformed into CPSP. That offers a new management goal in postoperative pain prevention.CT-guided hookwire localization have been proven to be benefical for VATS to diagnose and treat small pulmonary , it can shorten operation timing and increase surgery success rate. However, it causes roughly 23.8% severe pain and complaints included wire dislodgement, pneumothorax and haemorrhage during and after insertion. The question is whether or not the moderate-to-severe acute postoperative pain from hookwire localition will change the incidence and intensity of CPSP in VATS.

Nurses play a pivotal role in advanced practice, research, and education in the field of pain management. The pain management of hookwire localization may be a new vison in further research.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75
* patients who underwent underwent CT-guided localization before VATS
* ASA I-II
* BMI 18.5-30
* no serious complications after localization
* sign informed consent

Exclusion Criteria:

* could not complish underwent CT-guided localization
* selfexpression or visual dysfunction
* having emergency surgery
* a severe psychiatric illness
* having chronic pain problems in the chest area
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The institutional review board approved this prospective study. This study included 138 consecutive patients who underwent CT-guided localization before VATS , of which 69 using hookwire (Group A) and 69 without hookwire (Group B). The inclusion criteria were as follows: patients were planned to underwent VATS for lung cancer .
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
postoperative incidence and intensity of chronic pain after surgery | at postoperative 3rd month
  the incidence and severity（11-point numerical rating scale,0=painless, 10=woest pain）of pain was assessed after VATS operation
postoperative incidence and intensity of chronic pain after surgery | at postoperative 6th month
  the incidence and severity（11-point numerical rating scale, 0=painless, 10=worst pain）of pain was assessed after VATS operation

SECONDARY OUTCOMES:
postoperative length of stay in hospital | an average of 1 week
  the days between postoperative 1st day and day of discharge from hospital
satisfactory score | from the day discharge from hospital to postoperative 6th month
  Likert score (from 1 to 5),higher scores mean a better outcome
intensity of postoperative acute pain | from immediately after surgery(at postanesthesia care unit ) to postoperative 2nd day
  the severity(11-point numerical rating scale, 0=no pain, 10=worst pain) after VATS operation

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Department of Anesthesiology, Fudan University Shanghai Cancer Center;
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China